CLINICAL TRIAL: NCT07081152
Title: Long-term Iron Absorption and Losses in Young South African Women Living Without and With Overweight and Obesity
Brief Title: Iron Absorption and Losses in Young South African Women Living Without and With Overweight and Obesity
Acronym: RAYON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linda Malan (Other)
Collaborators: King's College London (Other); ETH Zurich (Switzerland) (Other)
Responsible Party: Sponsor-Investigator, Linda Malan, Prof, North-West University, South Africa
Organization: North-West University, South Africa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RAYON; 26891 (Other: International Atomic Energy Agency)
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Iron Deficiency; Inflammation
MeSH Terms: conditions — Obesity; Iron Deficiencies; Inflammation | interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Living without overweight/obesity (Active Comparator): Participants with body mass index between 18 and 24.9 kg/m2
  Interventions: Other: Ferrous sulfate
- Living with overweight/obesity (Experimental): Participants with body mass index equal to or greater than 28 kg/m2
  Interventions: Other: Ferrous sulfate

INTERVENTIONS:
Other: Ferrous sulfate — All participants will receive a single dose of 15 mg of iron as isotopically prepared ferrous sulfate labelled with 57Fe. The iron dose will be given with ascorbic acid to attain a molar ratio of ascorbic acid:iron of 2:1

SUMMARY:
Young women living with obesity (OB) have a greater risk of developing iron deficiency. Plus, the risk of anemia and/or ID in young women living with overweight (OW) and obesity (OB) is further increased by inadequate dietary intake and/or poor bioavailability of iron, as well as gastrointestinal and menstrual iron losses. It is not certain whether women living with OW/OB can meet their iron requirements from their day-to-day diet.

The aim of this study is to compare iron absorption and losses over a long period between women living with and without OW and OB. Secondary outcomes include iron and inflammation status, as well as dietary iron intake.

DETAILED DESCRIPTION:
Adiposity-related inflammation stimulates an increase in secretion of hepcidin hormone thus limiting the absorption of iron and increasing the risk for iron deficiency (ID). In addition, the risk of anemia and/or ID in young women living with overweight (OW) or obesity (OB) is further increased by inadequate dietary intake and/or poor bioavailability of iron, as well as gastrointestinal and menstrual iron losses. Although one study quantified iron losses and absorption in young African women using the stable isotope dilution method the focus was on normal-weight women. Thus, whether women living with OW/OB can meet their iron requirements from their habitual diet remains uncertain.

This is a longitudinal study including an iron absorption study (Phase 1) and a follow-up period (Phase 2) in women living with and without OW and OB.

In phase 1, 70 healthy, mildly- and non-anemic young women living with and without OW or OB will receive a test drink labelled with 15 mg of labelled ferrous sulfate (57Fe) (Visit 1). Fractional iron absorption from the test drink will be determined by measuring the incorporation of the isotopic label into red blood cells 14 days after administration (Visit 2), and will be compared between the two groups. Participants will then undergo a one-year equilibration period. During this time, they will be contacted monthly to ask about their health status, medication and supplements use, blood donation or transfusion, and whether they have fallen pregnant. About 1 year after isotope administration, participants will be contacted again and screened (Visit 3) for phase 2 of the study. Phase 2 of the study will involve 4 visits (Visits 4 to 7), where they will be followed up for 6 months. During this time, blood samples will be drawn every 8 weeks for the determination of isotopic composition. In addition, iron and inflammation status, as well as dietary intake of iron, including its absorption enhancers and inhibitors, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Of African descent
* BMI of 18.5 to 24.9 kg/m2 for participants living without OW/OB and BMI ≥ 28 kg/m2 for participants living with OW/OB
* Having low to moderate inflammation-adjusted iron stores (ferritin ≤50 µg/L)
* Absence of low-grade inflammation (CRP<2 mg/l) for participants living without OW/OB and presence of low-grade inflammation CRP 2-20 mg/l) for participants living with OW/OB
* Planning to reside in the study area for at least 2 years

Exclusion Criteria:

* Hemoglobin < 11 g/dl
* Treated or self-reported chronic or malabsorptive disorder
* Current use of chronic anti-inflammatory medication, like corticosteroids or non-steroidal anti-inflammatory medication
* Pregnancy or planning to become pregnant in the next 2 years
* Lactation
* Fear of needles or experiencing vaso-vagal episodes when exposed to blood
* Difficulty drawing blood due to poor quality veins
* Blood donation in the past 4 months or plans to donate blood during the study
* On a weight-loss diet or program or planning to start the same during the study
* Smoking
* Unwillingness to stop taking iron and /or vitamin C-containing supplements during phase 1 of the study

Additional inclusion criteria applicable to phase 2 of the study

* Labelled with stable iron isotope (tracer) for a minimum of one year
* Willingness not to start or stop contraceptive use during the 6 months
* BMI ≥ 18.5 to 24.9 kg/m2 for participants living without OW/OB and BMI ≥ 28 kg/m2 for participants living with OW/OB

Additional exclusion criteria applicable to phase 2 of the study

- Blood transfusion, intravenous iron infusion, blood donation or significant blood loss during the equilibration period

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Iron absorption | Visits 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Long-term iron absorption will be determined in, and compared between women living without and with OW/OB in Phase 2 of the study and will be proportional to the change in the concentration of iron isotope 57 in the erythrocyte over time.

SECONDARY OUTCOMES:
Iron losses | Visits 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Long-term iron losses will be determined in, and compared between women living without and with OW/OB in Phase 2 of the study and will be proportional to the change in the absolute amount of iron isotope 57 in the erythrocyte over time.
Iron balance | Visits 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Iron balance will be calculated in and compared between women living without and with OW/OB as the difference between iron absorption and iron losses.
Fractional iron absorption | Visit 2 (day 15)
  Fractional iron absorption from a single dose of 15 mg of isotopically-labeled iron will be compared between women living without and with OW/OB.
Iron status | Screening (Ferritin only), Visits 1 (day 1), 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Iron status will be determined by measuring plasma ferritin and soluble transferrin receptor.
Inflammation status | Screening (CRP only), Visit 1 (day 1), 3 (day 366;CRP only), 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Inflammation status will be determined by measuring plasma C-reactive protein (CRP) and alpha-1-acid glycoprotein.
  CRP will also be used to assess the absence or presence of low-grade inflammation at screening for phase 1 and visit 3, using a cut-off of <2 mg/l and 2-20 mg/l, respectively.
Dietary iron intake | Visits 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Dietary iron intake will be assessed using a quantified food frequency questionnaire.
Laboratory comparison of measurement of red blood cell isotope concentrations | Visit 2 (day 15), 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Iron isotope concentration measurements will be compared between the laboratories at North-West University and the Swiss Federal Institute of Technology Zurich.
Dietary intake of iron absorption enhancers | Visits 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Dietary intake of iron absorption enhancers like vitamin C will be determined using a quantified food frequency questionnaire.
Dietary intake of iron absorption inhibitors | Visits 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Dietary intake of iron absorption inhibitors like phytic acid will be determined using a quantified food frequency questionnaire.
Body fat percentage | Screening, Visits 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Body fat percentage will be assessed using the deuterium dilution technique and/or bioelectrical impedance analysis.
Waist circumference | Screening, Visits 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Waist circumference will be measured as an indicator of body fat distribution.
Hip circumference | Screening, Visits 4 (day 373), 5 (day 429), 6 (day 485) and 7 (day 541)
  Hip circumference will be measured as an indicator of body fat distribution.
Liver function | Screening
  Liver function will be assessed by measuring alanine transaminase and aspartate transaminase enzymes.
Gut inflammation | Screening
  Gut inflammation will be assessed by measuring gut integrity and inflammation biomarkers namely Intestinal fatty acid-binding protein (IFABP) and soluble cluster of differentiation 14 (sCD14).
Menstruation intensity | Day 373 to day 541
  Menstruation intensity will be assessed using a self-administered health diary
Haemoglobin | Screening
  Haemoglobin measurement will be compared between a point-of-care device (Hemocue) and an automated haematology analyser

CONTACTS AND LOCATIONS:
Overall Officials: Linda Malan, PhD, Principal Investigator — Centre of Excellence for Nutrition, North-West University; Mary Uyoga, PhD, Principal Investigator — Centre of Excellence for Nutrition, North-West University
Locations (1):
- Esté Vorster Research Facility, Potchefstroom, North West, South Africa